CLINICAL TRIAL: NCT03957811
Title: Intervention Project for Diabetic Foot Prevention Through the Development of a Vibratory Therapy Program at the National Rehabilitation Institute LGII
Brief Title: Effect of Whole-body Vibration on TcPO2
Acronym: WBV
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Rehabilitacion (Other Government)
Collaborators: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, Gerardo Rodríguez Reyes, Medical Science Researcher, Instituto Nacional de Rehabilitacion
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2416; 2234 (Other: Instituto Nacional de Ciencias Médicas y Nutrición)
Record Dates: First submitted 2019-05-17; First posted 2019-05-21 (Actual); Last update posted 2019-08-26 (Actual); Status verified 2019-08

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: There will be two parallel groups. One will receive the standard treatment for diabetes, and the other will receive standard treatment plus sessions of vibration exercise therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Controls (No Intervention): Subjects under treatment for diabetes will receive the standard treatment for their condition.
- Intervention (Experimental): Subjects under treatment for diabetes not diagnosed for diabetic foot will receive the standard treatment plus exercise on a vibrator platform for a period of 12 weeks.
  Interventions: Other: Whole body Vibration exercise

INTERVENTIONS:
Other: Whole body Vibration exercise — Intervention will consist of sessions of exercise on a whole body vibration platform, three times a week for 12 weeks.
  Arms: Intervention

SUMMARY:
In order to determine the effect of whole body vibration on TcPO2 levels in patients with type 2 diabetes, 40 subjects will undertake whole body vibration exercise three times a week for 12 weeks. TcPO2 will be measured before and after the intervention. A second control group with type 2 diabetes will also have TcPO2 levels measured before and after the 12 weeks of the study.

DETAILED DESCRIPTION:
Objective: To determine the effect of whole body vibration exercise on levels of TcPO2 measured in the feet of patients with type 2 diabetes, in order to create recommendations for prevention of diabetic foot.

Material and Methods: controlled open clinical trial consisting in 2 arms, as follows: 1) control group under care for type 2 diabetes, and 2) intervention group, who, in addition to the standard care, will undergo an exercise program of whole body vibration three times a week, with progressive intensity, for a period of 12 weeks. Partial pressure of transcutaneous oxygen (TcPO2) will be measured in the feet of the participants at baseline and after 12 weeks, with 40 patients per group.

Statistical analysis: demographic information of the subjects will be described as arithmetic means, standard deviation, percentages, frequencies. Comparison between groups will be done with Student t for independent data or Mann-Whitney U when convenient. Baseline and final measurements will be compared. inter and intra group comparisons will be made by repeated measurements. For qualitative values, chi square will be used. Multivariate analysis will be performed to control for confounding variables. The level of significance will be a value of 0.05.

ELIGIBILITY:
Inclusion Criteria:• Patients with diagnosis of type 2 diabetes less than or equal to six years, under care and having concluded the 4th or 5th medical visit.

* Non-smokers.
* Residents of Mexico City
* Both sexes.
* 40 to 69 years old.
* Agreeing to participate through signature of informed consent.
* HbA1c between 6.0 and 9.0 %.
* Blood pressure less than or equal to130/80.
* Total cholesterol ≤ 240 mg/dL, triglycerides ≤300 mg/dL.
* Stable weight over the last 6 months ( <10% variation).

Exclusion Criteria:• Patients with severe motor handicap and amputations of pelvic members.

* With exposed lesions in subcutaneous tissue (ulcers) in the sole of the foot, diabetic foot (Wagner 3 or more) or intermittent claudication.
* With important alterations in balance.
* With a recent surgery.
* Gravidity.
* Deep venous thrombosis.
* With pacemaker.
* Recent myocardial ischemia.
* Orthopedic implants.
* Recently-placed mammary prosthesis.
* Exoskeletal prosthesis.
* Discopathies.
* Neoplasia in the last 5 years.
* History of 2 episodes of severe hypoglycemia in the last year.
* Chronic kidney disease with creatinine clearance estimated at <60 ml/min.
* Severe non-proliferative retinopathy, uncontrolled macular edema.
* Hepatic failure (Child-Pugh "C") and/or heart failure (functional Class - NYHA-: III-IV).
* Patients with hemoglobinopathies, severe anemia (≤7.5 g/dL), known hemolytic disease.

Ages: 40 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-04-04 (Actual); Primary Completion 2019-12-20 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Effect of whole body vibration on TcPO2 levels | 12 weeks
  To know the effect of whole body vibration on TcPO2 levels measured in the foot in patients with type 2 diabetes

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Nacional de Rehabilitacion, Mexico City, Mexico City, Mexico